CLINICAL TRIAL: NCT07326462
Title: The Effects of Strength Training Volume, Intensity, and Breathing Techniques on Intraocular Pressure and Retinal Blood Vessels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: LithuanianSportsU-27
Record Dates: First submitted 2025-12-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
Keywords: intraocular pressure; exercise; Valsalva maneuver; retinal vessels
MeSH Terms: conditions — Motor Activity | interventions — Valsalva Maneuver

STUDY DESIGN:
Intervention Model Description: This is a crossover experimental study with 60 healthy adults, where each participant completes two exercise arms (isometric vs. isokinetic) under two breathing interventions (normal vs. Valsalva), separated by 2-3 days. The design allows controlled comparison of ocular and systemic responses to exercise and breathing techniques within the same individuals.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isokinetic exercise arm (Experimental): Protocol: Participants perform a 1-minute maximal voluntary isometric contraction of the knee extensors using a BIODEX dynamometer.
  Load setting: The maximum isometric load that each individual can sustain for 1 minute is determined during familiarisation. In the main session, participants work at 80% of their predetermined maximum load to avoid premature muscle failure.
  Nature of exercise: Static contraction (muscle generates force without changing length).
  Interventions: Diagnostic Test: Normal Breathing; Diagnostic Test: Valsalva maneuver
- Isometric exercise arm (Experimental): Protocol: Participants perform 1 minute of repeated isokinetic knee extensions and flexions at a controlled angular velocity on the BIODEX dynamometer.
  Velocity settings: Knee extension at 30°/s and knee flexion at 60°/s within the 0°-90° range of motion (0° = full extension).
  Nature of exercise: Dynamic contraction (muscle changes length while producing force against constant velocity resistance).
  Interventions: Diagnostic Test: Normal Breathing; Diagnostic Test: Valsalva maneuver

INTERVENTIONS:
Diagnostic Test: Normal Breathing — Participants perform the isometric or isokinetic exercise while following a controlled breathing rhythm:
  Inhale for 3 seconds
  Exhale for 3 seconds
  Breathing remains steady and continuous throughout the 1-minute exercise.
  Rationale: Represents a natural and safe breathing pattern during physical exertion, serves as the physiological baseline condition.
Diagnostic Test: Valsalva maneuver — Participants perform the same isometric or isokinetic exercise but finish the trial with a 10-second breath-hold at the end of the 1-minute exercise.
  This maneuver increases intrathoracic and intra-abdominal pressures, which are transmitted to ocular and vascular systems.
  Rationale: Common in athletic performance, but may cause significant intraocular pressure and retinal vascular fluctuations.

SUMMARY:
This study aims to determine the effects of different breathing patterns on ocular vasculature and intraocular pressure (IOP) during isokinetic and isometric strength exercises. It is hypothesized that higher ocular microcirculation changes and IOP values will be observed during the Valsalva maneuver compared to normal breathing in both exercise types. Additionally, ocular microcirculation and IOP changes are expected to be more pronounced during isometric exercises than during isokinetic exercises. The results will help establish optimal strength training strategies for both professional athletes and physically active individuals.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to evaluate the effects of different breathing patterns on ocular vasculature and intraocular pressure (IOP) during isokinetic and isometric strength exercise in healthy young adults.

The study protocol was approved by the Kaunas Regional Biomedical Research Ethics Committee, and all participants provided written informed consent prior to participation, in accordance with the Declaration of Helsinki.

Participants will attend experimental sessions during which ocular and cardiovascular parameters will be assessed before exercise, immediately after exercise, and during the recovery period.

Baseline assessments will include general anthropometric measurements and questionnaires related to physical activity and fatigue, as well as evaluation of ocular surface condition.

Retinal microcirculation will be assessed using non-mydriatic fundus photography, and intraocular pressure will be measured using a portable tonometry method. Blood pressure and oxygen saturation will also be monitored during study sessions.

Each participant will perform a standardized 1-minute strength exercise under two exercise modalities: isokinetic and isometric. A standardized warm-up will precede each exercise session.

Two breathing conditions will be evaluated during exercise: normal breathing and the Valsalva maneuver. The order of exercise modality and breathing condition will be randomized, and experimental sessions will be separated by an adequate washout period.

The planned sample size was determined a priori based on statistical power considerations to ensure adequate power to detect meaningful differences between study conditions.

Data will be analyzed using appropriate statistical methods. Descriptive statistics will be used to summarize study data. Normality of data distribution will be assessed, and non-parametric methods will be applied when appropriate. Repeated-measures and between-condition comparisons will be conducted, with adjustments for multiple comparisons applied as needed. Statistical significance will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18-40 years old
2. Peak IOP <21 mmHg in the modified DTC
3. Open angle at gonioscopy
4. Optic disc with cup-to-disc ratio <0.6 with no signs of glaucomatous neuropathy
5. Not currently taking any medication
6. Non-smokers, no physical and mental disabilities
7. Blood pressure up 120/80 mmHg and heart rate (HR) 60-90 rpm at rest
8. BMI (18.5-34.8) kg/m2

Exclusion Criteria:

1. Presence of any ocular disease (with the exception of refractive errors)
2. Anxiety or depressive disorders
3. History of ocular trauma or surgery
4. Pregnancy
5. Use of any kind of oral/topical steroids
6. Any diagnosed chronic health condition such as cardiovascular disease including hypertension and or previous physical injuries that could impact their safe participation
7. Evidence of ocular pathology due to narrow anterior chamber angles, elevated IOP greater than or equal to 21mm Hg, optic nerve or retinal pathology, cup: disc ratio of greater than 0.6 or asymmetry of cup: disc ratio of greater than 0. 2.
8. Refractive error more than ±4.00 diopters, astigmatism greater than 3.00 diopters.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
1. Intraocular Pressure (IOP) | 3 days
  Tool: Icare portable tonometer (Icare, Tiolat Oy, Helsinki, Finland).
  Description: Measures the pressure inside the eye, caused by the aqueous humor pressing against the eye wall.
  Rationale: IOP is a key factor in glaucoma development and progression. Monitoring fluctuations during exercise and different breathing techniques is critical.
  Timing: Baseline (before exercise), immediately post-exercise, and at 5, 10, 15 minutes after exercise.
2. Retinal Microcirculation | 3 days
  Tool: Aurora handheld non-mydriatic fundus camera (Optomed, Finland).
  Description: Digital fundus photography to measure retinal vessel diameters (arterioles and venules) in the superior and inferior temporal quadrants, near the optic disc margin.
  Rationale: Retinal vessel diameter is a biomarker for cardiovascular health and provides insights into ocular blood flow changes during stress.
  Timing: Same schedule as IOP (before, immediately after, and 5, 10, 15 minutes post-exercise).
3. Blood pressure (BP) | 3 days
  Tool: Omron BP742N automatic arm blood pressure monitor (Omron Healthcare, Japan).
  Description: Monitors systolic and diastolic blood pressure levels.
  Rationale: To capture systemic cardiovascular responses during isometric vs. isokinetic exercise and different breathing conditions.
  Timing: Baseline, immediately after, 5, 10, and 15 minutes post-exercise.
4. Oxygen Saturation (SpO₂) | 3 days
  Tool: Pulse oximeter (Omron).
  Description: Monitors peripheral blood oxygen levels.
  Rationale: Evaluates systemic oxygen delivery and breathing effects (especially relevant with Valsalva maneuver).
  Timing: During the exercise protocol (exact points not deeply detailed in file but implied to match BP).
5. Eye Dryness | 3 days
  Tool: Schirmer Test (TearFlo strips).
  Description: Filter paper strips placed inside the lower eyelid for 5 minutes; length of wetting indicates tear production.
  Rationale: Assesses ocular surface health, as exercise and breathing methods may influence tear production and comfort.
  Timing: At baseline (before experimental trials).
6. Anthropometric Data | 3 days
  Tools:
  Leicester Height Metre for height.
  Tanita TBF-300 body composition scale for weight and body fat %.
  Derived Measurement: Body Mass Index (BMI = weight/height²).
  Rationale: Provides participant characteristics for standardization and analysis.
Questionaire no. 1 | 3 days
  Validated Baecke questionnaire → Physical activity level. Rationale: Captures subjective perception of workload alongside physiological measures.
Questionnaire no.2 | 3 days
  Fatigue assessment questionnaires → Subjective fatigue. Rationale: Captures subjective perception of fatigue alongside physiological measures.
Questionnaire no. 3 | 3 days
  Rating of Perceived Exertion (RPE) → Subjective exercise intensity. Rationale: Captures subjective perception of exertion alongside physiological measures.

CONTACTS AND LOCATIONS:
Overall Officials: Vytautas Streckis, phD, Prof., Study Director — Lithuanian Sports University